CLINICAL TRIAL: NCT05230082
Title: Acupuncture Treatment for Individuals With Myasthenia Gravis
Brief Title: Acupuncture in Myasthenia Gravis (AcuMG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A21-197
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start (Experimental): Patients will receive acupuncture treatment two times per week for 12 weeks.
  Interventions: Other: Acupuncture
- Delayed start (Active Comparator): Patients will act as control group for the first 12 weeks then will receive acupuncture treatment two times per week for 12 weeks.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.

SUMMARY:
The purpose of the study is to determine the effect acupuncture treatment on individuals with a diagnosis of Myasthenia Gravis (MG). A total of 20 people with MG will be enrolled in this study to receive acupuncture treatment 2 times a week for 12 weeks. Participants will be randomized into two groups: 1) Immediate start and 2) Delayed start (12 weeks). The delayed start group will act as a control group for the first 12 weeks, but then receive acupuncture treatment for 12 weeks. It is hypothesized that patients with MG who receive acupuncture treatment will have improved quality of life and activities of daily living compared to no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide and provision of signed and dated informed consent form
* Age 18-80
* Diagnosis of MG

Exclusion Criteria:

* Non-English speaking
* Participation in acupuncture treatment outside of the study, while enrolled
* History of any other serious neurological, psychiatric, chronic pain disorders, or seizures
* History of bleeding diathesis, other bleeding disorders, or syncope with needle puncture
* History of cardiac arrhythmia or current pacemaker, neurostimulator, or other implanted stimulation device
* Recent or active substance use disorder
* Women who are currently pregnant, lactating, or planning to become pregnant during the study
* Any other medical conditions that could affect their ability to participate in acupuncture treatments for the study duration (as determined by study investigators)
* Active participation or past participation ≤3 months in any other interventional study.
* Unwilling to participate in all study related activities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda A Herrmann, PhD, Principal Investigator — HealthPartners Neuroscience Research; Gaurav K Guliani, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Start: Patients will receive acupuncture treatment two times per week for 12 weeks.
  Acupuncture: Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.
  Period 1: Acupuncture - Weeks 1-12 Period 2: No Acupuncture - Weeks 13-27
- Delayed Start: Patients will act as control group for the first 12 weeks then will receive acupuncture treatment two times per week for 12 weeks.
  Acupuncture: Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.
  Period 1: No Acupuncture - Weeks 1-12 Period 2: Acupuncture - Weeks 13-24
Period: Period 1: Weeks 1-12
Arm/Group | Immediate Start | Delayed Start
Started | 10 | 14
Completed | 6 | 13
Not Completed | 4 | 1
Period: Period 2: Weeks 13-24
Arm/Group | Immediate Start | Delayed Start
Started | 6 | 13
Completed | 6 | 11
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Start | Delayed Start | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 59 (13) | 62 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Time since MG Diagnosis [Mean (Standard Deviation); unit: years] | 6 (8) | 10 (11) | 8 (9)
Diagnosis Classification [Count of Participants; unit: Participants] — A base treatment of 21 needling points was used for all study participants. An unscored symptom severity scale was developed to help examine individual symptoms. Acupuncturists made a differential diagnosis to determine the diagnostic categories that were used to classify patterns of disharmony or imbalance within the body. Up to 9 additional points could be added to the base treatment, allowing for individual treatment.
  Yin - nourishment and repair functions Yang - defense and immune functions Stagnation pronounced - disruption in the flow of Qi (energy) and blood, often marked by pain.
  Participants
    Yang deficiency | 4 | 5 | 9
    Yin deficiency | 2 | 4 | 6
    Stagnation pronounced | 1 | 3 | 4
    Base treatment | 1 | 0 | 1
    Withdrawn before classification | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Effect of Acupuncture on Quality of Life in Patients With MG
Description: A brief 15-item disease specific questionnaire. Myasthenia gravis-quality of life 15 (MG-QOL15). A higher score indicates a lower quality of life.[range: 0-30]
Time Frame: pre-acupuncture treatment and post-acupuncture treatment
Population: Participants withdrew prior to the post-treatment measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 10 | 14
score on a scale
  pre-treatment | 10.8 (6.7) | 9.4 (7.4)
  post-treatment: number analyzed (Participants) | 7 | 12
  post-treatment | 3.6 (2.0) | 8.3 (7.0)

2. Secondary Outcome: To Determine the Effect of Acupuncture on Activities of Daily Living in Patients With MG
Description: A brief 8-item disease specific questionnaire. Myasthenia gravis-activities of daily living (MG-ADL). A higher score indicates activities of daily living are more difficult.[range: 0-24]
Time Frame: pre-acupuncture treatment and post-acupuncture treatment
Population: Participants withdrew prior to the post-treatment measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 10 | 14
score on a scale
  Pre-treatment | 5.0 (3.1) | 3.6 (3.0)
  Post-treatment: number analyzed (Participants) | 7 | 12
  Post-treatment | 2.3 (1.6) | 3.5 (2.4)

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- Immediate Start - Period 1 - Acupuncture Treatment; Immediate Start - Period 2 - No Intervention: Patients will receive acupuncture treatment two times per week for 12 weeks.
  Acupuncture: Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.
- Delayed Start - Period 1 - No Intervention; Delayed Start - Period 2 - Acupuncture Treatment: Patients will act as control group for the first 12 weeks then will receive acupuncture treatment two times per week for 12 weeks.
  Acupuncture: Acupuncture treatments will be separated by a minimum of two days and a maximum of 14 days. Treatment sessions will be identical for both groups. Standard, sterile stainless-steel, disposable needles will be inserted at acupuncture points with a total of 18 needles for each treatment session. The depth of the needle will be approximately 10-20 millimeters. Needles will be left in place for 30 minutes.
Arm/Group | Immediate Start - Period 1 - Acupuncture Treatment | Immediate Start - Period 2 - No Intervention | Delayed Start - Period 1 - No Intervention | Delayed Start - Period 2 - Acupuncture Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/10 | 1/10 | 8/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Period 1 - Acupuncture Treatment (N=10) | Immediate Start - Period 2 - No Intervention (N=10) | Delayed Start - Period 1 - No Intervention (N=14) | Delayed Start - Period 2 - Acupuncture Treatment (N=14)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | NA | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Period 1 - Acupuncture Treatment (N=10) | Immediate Start - Period 2 - No Intervention (N=10) | Delayed Start - Period 1 - No Intervention (N=14) | Delayed Start - Period 2 - Acupuncture Treatment (N=14)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 1 (1) | 1 (2) | NA
Needling pain/bruising (Injury, poisoning and procedural complications) | 3 (5) | 0 (0) | 3 (4) | NA
Headache (General disorders) | 1 (4) | 0 (0) | 2 (2) | NA
Sinus issues (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0) | NA
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2) | NA
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | NA
Sleep disturbances (General disorders) | 0 (0) | 0 (0) | 2 (2) | NA
COVID-19 (General disorders) | 0 (0) | 0 (0) | 2 (2) | NA
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | NA
Eye Tearing (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Vaccine Reactions (General disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Eye Ptosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Hip Vibration Sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Restless Leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Phantom Sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Muscle Numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Eye Bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Pneumonia and Flu (General disorders) | 1 (1) | 0 (0) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05230082/Prot_SAP_000.pdf